CLINICAL TRIAL: NCT04458220
Title: Research on Early Warning and Solution System of Difficult Airway in Perioperative Period Based on Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2020-T233-1
Record Dates: First submitted 2020-06-18; First posted 2020-07-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Difficult Airway

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult airway: C-L≥Ⅲ grade
  Interventions: Other: photo and voice obtained
- none difficult airway: C-L<Ⅲgrade
  Interventions: Other: photo and voice obtained

INTERVENTIONS:
Other: photo and voice obtained — The 3D face scanner and camera is used to obtain 3D or 2-dimensional portrait images of patients in different positions and from different angles.The Hi-Fi Recorder is used to obtain sound samples of patients in different word.

SUMMARY:
The study is performed in Shanghai Ninth People's Hospital Affiliated with Shanghai Jiao Tong University School of Medicine . According to inclusion and exclusion criteria ,the investigators are expected to enroll 16000 participants who performed endotracheal intubation under general anesthesia. All enrolled participants must sign a written informed consent.In the preset studio,The 3D face scanner and camera is used to obtain 3D or 2-dimensional portrait images of patients in different positions and from different angles.The Hi-Fi Recorder is used to obtain sound samples of patients in different word.Then,Statistical experts use quantitative software to quantify the data.The investigators will put all the data and images into a confidential database in order to build a large database of difficult airways.

Anesthesiologist will give every patient an endotracheal intubation as planned. After that the anesthesiologist will be asked to fill out the questionnaire immediately.This questionnaire allows obtaining a ground truth for the intubation difficulty.All data will be used for AI deep learning and intelligent analysis,Several of the most relevant landmarks will be selected to build an early warning model.The overall study did not involve any intervention in the process of anaesthesia and operation of the patients, only the three-dimensional facial images of the patients were obtained, without any trauma or injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be intubated under general anesthesia.

Exclusion Criteria:

* Patients with deaf-mutism or communication disorders.
* Patients with language deficiency or non-native language.
* Patients with mental or central nervous system disease.
* Patients with stupefaction or disturbance of consciousness.
* Patients with terrible injury.
* Patients cannot follow instructions to perform standard actions.
* Patients participated in other relevant clinical investigation in the past 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study is performed in Shanghai Ninth People's Hospital Affiliated with Shanghai Jiao Tong University School of Medicine . According to inclusion and exclusion criteria ,We are expected to enroll 16000 participants who performed endotracheal intubation under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosed as a difficult airway | Just after intubation
  C-L≥Ⅲ grade

SECONDARY OUTCOMES:
Difficult mask ventilation | 2 minutes after administration of Rocuronium
  The difficult mask ventilation was defined as follows: (1) the inability of an unassisted anesthesiologist to maintain oxygen saturation, as measured by SpO2<92% with 100% oxygen and positive-pressure mask ventilation; (2) significant gas flow leakage around the face mask; (3) the need to increase the gas flow to more than 15 L/min and use the oxygen flush valve more than twice (4) absence of visible chest movement; (5) the necessity to switch to a two-handed mask ventilation technique; (6) the need for operator substitution or addition.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, Dr, Study Chair — The Ninth People's Hospital of Shanghai Jiaotong University School of Medicine
Locations (1):
- The Ninth People's Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04458220/ICF_000.pdf